CLINICAL TRIAL: NCT06017518
Title: An Observational Study of Local Relapse After High Grade Osteosarcoma
Acronym: OSTEO LR
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: OSTEO LR
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
multicenter retrospective and prospective study in patients with high-grade osteosarcoma

DETAILED DESCRIPTION:
This is a multicenter retrospective and prospective study that will analyze all cases with of diagnosis of local relapse in high-grade osteosarcoma from 01 January 1980 and all new cases referring to each participant site.

ELIGIBILITY:
Inclusion Criteria:

* Patients who experienced LR as first event of recurrence after treatment for localized high-grade osteosarcoma of bone, including cases with synchronous lung metastases
* Adequate patient compliance to follow-up visits
* Written informed consent prior to any study-specific analysis and/or data collection
* No age limits

Exclusion Criteria:

* Cases of LR demonstrated after > 3 months after metastatic disease
* Impossibility to ensure adequate compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who experienced local relapse as first event of recurrence after treatment for localized high-grade osteosarcoma of bone, including cases with synchronous lung metastases
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
post local relapse survival | 24 months follow up
  the aim of the study is to analyse the factors influencing post local relapse survival

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna, BO
  - Azienda Ospedaliero-Universitaria Pisana, Pisa, PI

DOCUMENTS (1):
  • Study Protocol (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT06017518/Prot_000.pdf